CLINICAL TRIAL: NCT04130087
Title: The Effects of a Single Dose on Reward and Emotional Processing in Healthy Volunteers
Brief Title: Selegiline and Reward Processing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R64689/RE001
Record Dates: First submitted 2019-09-24; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: Reward; Selegiline; Cognition
MeSH Terms: interventions — Selegiline

STUDY DESIGN:
Intervention Model Description: Placebo controlled trial.
  27 participants will be allocated to receive a single 10mg of selegiline and the same number will receive a single dose of placebo (lactose tablet.)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomisation code will be drawn up by a researcher not involved in the study using a randomisation tool online (https://www.sealedenvelope.com/simple-randomiser/v1/lists). The study randomisation code will be kept in a sealed envelope in a dedicated cabinet in Neurosciences Building of The Department of Psychiatry. At the end of the study, the randomisation blind will be broken by the principal investigator by opening the randomisation code envelope.
  Blinding will be achieved by identical encapsulation of the selegiline and the placebo using the Departmental Standard Operating Procedure for drug encapsulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selegiline Group (Experimental): 27 healthy participants who will be administered a single 10mg tablet of selegiline hydrochloride.
  Interventions: Drug: Selegiline Hydrochloride 10 MG
- Placebo Group (Placebo Comparator): 27 healthy participants who will be administered a single lactose tablet (placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selegiline Hydrochloride 10 MG — Single 10mg tablet of Selegiline Hydrochloride
  Arms: Selegiline Group
Drug: Placebo — Single Placebo Tablet, identical appearance to experimental tablet.
  Arms: Placebo Group

SUMMARY:
There has been growing interest in the relationship between reward processing and clinical symptoms of depression such as anhedonia (loss of interest and response to pleasurable activities).

The aim of the study is to investigate the acute effects of a single dose of selegiline (an irreversible monoamine oxidase B inhibitor) on reward and emotional processing in healthy volunteers.

DETAILED DESCRIPTION:
There has been growing interest in the relationship between reward processing and clinical symptoms of depression such as anhedonia (loss of interest and response to pleasurable activities). Studies in animals have suggested that the neurotransmitter, dopamine, plays a key role in reward processing. This has given rise to the suggestion that in depression, decrements in dopamine activity lead to impaired reward processing which cause symptoms such as anhedonia and low motivation.

Research in humans into dopamine and reward is limited by suitable pharmacological means to manipulate dopamine activity safely and effectively.

To our knowledge, no previous research has studied the effects of acute administration of the licensed drug, selegiline, on reward and emotional processing. However, a single dose of selegiline effectively inhibits monoamine oxidase B (MAO-B), which should lead to increased dopamine availability in the CNS. Therefore, selegiline may be a useful tool to explore the effect of modifying dopamine availability on reward processing. Acquiring such knowledge through this study could assist in the clinical use of MAO-B inhibition as a target to ameliorate symptoms such as anhedonia as well as increasing our general understanding of reward processing in healthy individuals.

The aim of this study is to explore the effects of acute administration of a standard (10mg) dose of selegiline on reward and emotional processing versus a placebo, in healthy volunteers. At this dose selegiline only has an -MAO-B function therefore the specific impact of MAO-B blockade on reward and emotional processing can be explored.

Research Question: What effect will the administration of a single dose of selegiline have on reward and emotional processing in healthy volunteers?

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age
* Able to give informed consent for study participation
* Sufficient fluency in English to understand and complete the neuropsychological tasks

Exclusion Criteria:

* Current usage of other regular medication (including the contraceptive pill, the Depo-Provera injection or the progesterone implant, and hormone replacement therapy)
* Any past or current Axis 1 DSM-IV psychiatric disorder
* Significant medical condition
* Pulse < 60 beats per minute at baseline screening
* Current or past gastro-intestinal disorder or irritable bowel syndrome
* Current pregnancy or breastfeeding
* Known lactate deficiency or any other problem absorbing lactose, galactose or glucose
* Current or past history of drug or alcohol dependency
* Participation in a psychological or medical study involving the use of medication within the last 3 months
* Previous participation in a study using the same, or similar, emotional processing tasks
* Smoker > 5 cigarettes per day
* Typically drinks > 6 caffeinated drinks per day

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-09-10 (Estimated); Study Completion 2020-09-10 (Estimated)

PRIMARY OUTCOMES:
Total monetary amount won in reward learning task. | Tested one hour after selegiline/placebo ingestion
  During this task participants have to repeatedly choose between 2 options. On each trial one of the options, if chosen by the participant, will result in the participant winning money. The participant simply has to learn which is the best option to choose so as to win as much money as possible.
Reaction times (milliseconds) in reward learning task | Tested one hour after selegiline/placebo ingestion
  During this task participants have to repeatedly choose between 2 options. On each trial one of the options, if chosen by the participant, will result in the participant winning money. The participant simply has to learn which is the best option to choose so as to win as much money as possible.
Reward sensitivity in reward learning task | Tested one hour after selegiline/placebo ingestion
  During this task participants have to repeatedly choose between 2 options. On each trial one of the options, if chosen by the participant, will result in the participant winning money. The participant simply has to learn which is the best option to choose so as to win as much money as possible.

SECONDARY OUTCOMES:
Reaction Time (milliseconds) on the Faces Dot Probe Task (FDOT) | Tested one hour after selegiline/placebo ingestion
  The FDOT assesses attention to positive versus negative stimuli using a reaction time measure. Two faces are presented vertically on the computer screen and replaced by a pair of dots, to which the participant has to respond by indicating whether the dots are vertically or horizontally aligned. On some trials, one of the two faces presented has an emotional expression (fearful or happy). On half of the trials, the faces are presented very briefly and immediately replaced by a jumbled face mask. The reaction time to respond to the dots can be used as a measure of attention to the emotional faces.
Reaction time (milliseconds) in an Emotional Categorisation Task (ECAT) | Tested one hour after selegiline/placebo ingestion
  The ECAT assesses speed to respond to positive and negative self-referent personality descriptors. Sixty personality characteristics (30 per valence) selected to be disagreeable (eg, sneering, untidy, hostile) or agreeable (eg, cheerful, honest, optimistic) are presented. The participants are asked whether they would like or dislike to be referred to as each characteristic.
Performance (number of words recalled) in an emotional recall task (EREC) | Tested one hour after selegiline/placebo ingestion
  The EREC is a surprise free recall task to assess the incidental encoding of emotional stimuli. Participants are asked to recall as many of the words previously presented in the ECAT task (See Outcome Measure 4) as they can. The relative recall of positive versus negative words gives a measure of emotional biases in memory. This task is not computerised - participants write the recalled words on paper.
Percentage Accuracy(%) on facial expression recognition task (FERT) | Tested one hour after selegiline/placebo ingestion
  The FERT assesses the interpretation of facial expressions. Faces with seven different basic emotions (happiness, fear, anger, disgust, sadness, surprise, neutral) are displayed on the screen and participants are required to indicate the expression on the face via a button-press. Different intensity levels of each emotion are presented, which increases the ambiguity of the facial expression and the sensitivity of the task.
Reaction times (milliseconds) on facial expression recognition task (FERT) | Tested one hour after selegiline/placebo ingestion
  The FERT assesses the interpretation of facial expressions. Faces with seven different basic emotions (happiness, fear, anger, disgust, sadness, surprise, neutral) are displayed on the screen and participants are required to indicate the expression on the face via a button-press. Different intensity levels of each emotion are presented, which increases the ambiguity of the facial expression and the sensitivity of the task.
Percentage accuracy (%) in an Emotional Recognition Memory Task (EMEM) | Tested one hour after selegiline/placebo ingestion
  The EMEM measures recognition memory for affective words. Participants are presented with a series of words comprising the pleasant and unpleasant personality words that were previously presented to them in the ECAT, and a set of previously unseen distracter words. For each word, participants are required to report whether they have previously seen the word.
Reaction times (milliseconds) in Emotional Recognition Memory Task (EMEM) | Tested one hour after selegiline/placebo ingestion
  The EMEM measures recognition memory for affective words. Participants are presented with a series of words comprising the pleasant and unpleasant personality words that were previously presented to them in the ECAT, and a set of previously unseen distracter words. For each word, participants are required to report whether they have previously seen the word.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Harmer, PhD, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Vrieze E, Pizzagalli DA, Demyttenaere K, Hompes T, Sienaert P, de Boer P, Schmidt M, Claes S. Reduced reward learning predicts outcome in major depressive disorder. Biol Psychiatry. 2013 Apr 1;73(7):639-45. doi: 10.1016/j.biopsych.2012.10.014. Epub 2012 Dec 8. PMID 23228328
- [Background] Admon R, Pizzagalli DA. Dysfunctional Reward Processing in Depression. Curr Opin Psychol. 2015 Aug 1;4:114-118. doi: 10.1016/j.copsyc.2014.12.011. PMID 26258159
- [Background] Krystal JH, Sanacora G, Duman RS. Rapid-acting glutamatergic antidepressants: the path to ketamine and beyond. Biol Psychiatry. 2013 Jun 15;73(12):1133-41. doi: 10.1016/j.biopsych.2013.03.026. PMID 23726151
- [Background] Machado-Vieira R, Salvadore G, Diazgranados N, Zarate CA Jr. Ketamine and the next generation of antidepressants with a rapid onset of action. Pharmacol Ther. 2009 Aug;123(2):143-50. doi: 10.1016/j.pharmthera.2009.02.010. Epub 2009 May 3. PMID 19397926
- [Background] Heinonen EH, Anttila MI, Nyman LM, Pyykko KA, Vuorinen JA, Lammintausta RA. Inhibition of platelet monoamine oxidase type B by selegiline. J Clin Pharmacol. 1997 Jul;37(7):597-601. doi: 10.1002/j.1552-4604.1997.tb04341.x. PMID 9243352